CLINICAL TRIAL: NCT03539341
Title: Randomized Controlled Trial of an Evidence-informed Parenting Intervention to Prevent Violence Against Young Children by Parents and Primary Caregivers in Thailand
Brief Title: Parenting for Lifelong Health - Thailand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Bureau of Inspection, Ministry of Public Health (Unknown); Regional Health Center 8 in Udon Thani (Unknown); Udon Thani Regional Hospital (Unknown); Boromarajonani College of Nursing (Ministry of Public Health) (Unknown); United Nations Children's Fund (UNICEF) Thailand (Unknown); Mahidol Oxford Tropical Medicine Research Unit (Other); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HCR17011
Record Dates: First submitted 2018-04-27; First posted 2018-05-29 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Parent Child Abuse; Domestic Violence; Child Behavior Problem; Child Neglect; Depression, Anxiety; Parent-Child Relations; Parenting; Parent-child Problem
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study will use a randomised controlled trial design to test the effects of the Parenting for Lifelong Health 2-9 Thailand programme in comparison to participants allocated to receiving care as usual in the control group (N = 120 parents and primary caregivers of children ages 2 to 9 years; 1:1 intervention to control group ratio).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLH-Thailand parenting programme (Experimental): Trained facilitators and coaches will deliver the programme over eight weekly sessions at the Udon Thani Regional Hospital during the feasibility pilot and the RCT. During the RCT, the 60 parents/primary caregivers in the intervention group will be divided into 4 groups of 15 participants, with each group overseen by 2 facilitators and 1 coach. Core session activities may include discussion about assigned home activities, core parenting principles, illustrated stories, role-plays, and problem solving. Home visits will be conducted by facilitators to those parents/primary caregivers who miss sessions or require additional support, and SMS/LINE messages will be delivered to all participants twice per week with relevant parenting tips and reminders to attend the upcoming session.
  Interventions: Behavioral: PLH-Thailand parenting programme
- Control (care as usual) (Other): The control will be an inactive condition of standard care at the time of the intervention. 'Standard care' may include access to Parent Schools in Mother and Child Health clinics at public hospitals, which are provided in some provinces and districts in Thailand. The delivery of services at Parent Schools are guided by the Ministry of Public Health Handbook for Parent Schools, which appear to be open to adaptation at the local level. At Parent Schools, three to five sessions are provided to parents in groups or one-on-one by hospital health personnel.
  Interventions: Other: Control (care as usual)

INTERVENTIONS:
Behavioral: PLH-Thailand parenting programme — Parenting programmes include developing positive caregiver-child interaction through child-led play and emotional communication, praise and rewards to encourage positive child behaviour, limit-setting behaviours such as effective instruction giving and establishing consistent household rules, and non-violent discipline strategies to replace harsh parenting and corporal punishment.
  Arms: PLH-Thailand parenting programme
Other: Control (care as usual) — The control will be an inactive condition of standard care at the time of the intervention. 'Standard care' may include access to Parent Schools in Mother and Child Health clinics at public hospitals, which are provided in some provinces and districts in Thailand.
  Arms: Control (care as usual)

SUMMARY:
Pilot design:

The feasibility pilot of PLH for Young Children in Thailand has a single-site, pre-post design with no control group, with the aims of assessing programme implementation, cultural and contextual relevance, and study feasibility. Although there is no comparison group and it is not designed to test effects, the pilot also has a provisional goal of reductions in child physical and emotional abuse at one-month post-intervention.

RCT design:

The RCT of PLH for Young Children Thailand is a randomized, controlled, observer-blinded, single-site trial with two parallel groups and a primary endpoint goal of reductions in child physical and emotional abuse at one month and three-months post-intervention. Randomisation will be performed at the individual level with a 1:1 allocation ratio.

Allocation: Using a 1:1 allocation ratio, the 120 participants will be randomly assigned to either the intervention or control group using the concealed computerized programme Sealed Envelope. An external researcher based at the Department of Social Policy and Intervention at the University of Oxford, and who is not directly involved in the study, will generate the random sequence. The Project Coordinator and Co-Investigator McCoy will notify participants of their allocation status via telephone following the collection of baseline data, in order to ensure that participants remain blind to their status during the initial assessment.

Blinding: Due to the involvement of facilitators and coaches in the delivery of the programme, blinding will not be possible for deliverers; moreover, participants cannot be blinded to their allocation status following the initial assessment. However, the allocation status of other participants will be kept concealed from participants in order to reduce the risk of contamination. Data collectors gathering outcome and process evaluation data, as well as statisticians providing support in data analysis, will be blinded to participant allocation status for the purposes of minimizing assessment bias. Cases of compromised blinding will be immediately reported to the Research Manager, who will consult with the research team on an appropriate course of action. Un-blinding of participants will only be permitted if any instances of significant harm due to participation in the study are reported by a participant or any member of the project team at any stage of the study.

This study is funded by the United Nations Children's Fund (UNICEF) Thailand and the Department of Social Policy and Intervention, University of Oxford.

UNICEF grant reference: PCA/THLC/2017/002

ELIGIBILITY:
Adult inclusion criteria:

1. Men or women aged 18 or older;
2. Serves as the primary caregiver of a child in the household between the ages of 2 and 9;
3. Parent passes the screening interview, based on the Multiple Indicator Cluster Survey (MICS) version 6 module on child discipline;
4. Provides consent to participate in the full study; and
5. Agrees to participate in the PLH for Young Children Thailand parenting programme.

Child inclusion criteria:

1. Aged 2 to 9 years; and
2. Parent/primary caregiver meets the above inclusion criteria.

Inclusion criteria for programme facilitators, who will deliver the PLH for Young Children Thailand programme:

1. Age 18 or older;
2. Prior participation in a five-day facilitator training workshop provided by PLH Trainers; and
3. Agreement to deliver the entire eight session PLH for Young Children Thailand programme.

Adult exclusion criteria:

1. Any adult exhibiting severe mental health problems or acute mental disabilities;
2. Any adult who is unavailable for participation in the PLH for Young Children Thailand programme at time of recruitment;
3. Any adult who has already participated in the feasibility pilot.

Child exclusion criteria:

Any child exhibiting acute physical or mental disabilities.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Change in frequency of child maltreatment (physical and emotional abuse) | Differences between groups at T2 (4 months) and T3 (7 months)
  Child maltreatment: physical & emotional abuse (self-report)
  Physical abuse (including abusive discipline) and emotional abuse will be measured using 20 items from an adapted and expanded version of the International Society for the Prevention of Child Abuse and Neglect (ISPCAN) Child Abuse Screening Tool-Trial Caregiver version (ICAST-T). The ICAST-T measures parental reports of the incidence of abuse perpetrated against their child over the past month using a frequency score on a scale of 0 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did you discipline [Child Nickname] by pushing, grabbing, or kicking him/her?"). This study will assess overall indication of previous child abuse (0 = no abuse; 1 = previous abuse), and frequency of overall abuse by summing all of the subscales. An indication of previous child abuse and a higher frequency of overall abuse represents a worse outcome.

SECONDARY OUTCOMES:
Change in frequency of physical and emotional abuse | Differences between groups at T2 (4 months) and T3 (7 months)
  Child maltreatment: physical and emotional abuse (self-report)
  Physical abuse (including abusive discipline) and emotional abuse will be measured using 20 items from an adapted and expanded version of the International Society for the Prevention of Child Abuse and Neglect (ISPCAN) Child Abuse Screening Tool-Trial Caregiver version (ICAST-T). The ICAST-T is an adaptation of the multi-national and consensus-based survey instrument ICAST-Parent version (ICAST-P), which has been used successfully in low and middle-income countries. The ICAST-T measures parental reports of the incidence of abuse perpetrated against their child over the past month using a frequency score on a scale of 0 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did you discipline [Child Nickname] by pushing, grabbing, or kicking him/her?"). This study will assess incidence of child maltreatment for physical abuse (13 items) and emotional abuse (7 items) by summing each individual subscale.
Change in number of instances of physical and emotional abuse | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Child maltreatment (physical and emotional abuse) will also be measured through the Home Observation for Measurement of the Environment (HOME) Inventory - Abusive and Harsh sub-scale. The original HOME Early Childhood and Middle Childhood Inventory Forms will be discussed and finalized by the Parenting Experts Working Group during the formative evaluation. The Abusive and Harsh sub-scale is expected to contain six items that utilize dichotomous scoring, with two items assessed via interview in the home regarding whether the parent used physical punishment or yelled at the child during the past week, and four items assessed via observation regarding whether the parent scolded or yelled; used physical restraint; hit, slapped, spanked, or kicked; and pushed, pulled, or pinched the child during the home visit.
Change in frequency of child maltreatment (physical and emotional abuse) | Differences between groups at T2 (4 months), controlling for T1 (baseline).
  Child maltreatment: physical & emotional abuse (self-report)
  Physical abuse (including abusive discipline) and emotional abuse will be measured using 20 items from an adapted and expanded version of the International Society for the Prevention of Child Abuse and Neglect (ISPCAN) Child Abuse Screening Tool-Trial Caregiver version (ICAST-T). The ICAST-T measures parental reports of the incidence of abuse perpetrated against their child over the past month using a frequency score on a scale of 0 to 7, or 8 or more times (e.g., "In the past 4 weeks, how often did you discipline [Child Nickname] by pushing, grabbing, or kicking him/her?"). This study will assess overall indication of previous child abuse (0 = no abuse; 1 = previous abuse), and frequency of overall abuse by summing all of the subscales.
Change in frequency of positive parenting | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Positive parenting behaviours will be assessed using the Parenting Young Children Scale (PARYC) (21 items), which measures the frequency of positive parenting (7 items), setting limits (7 items) and proactive parenting (7 items) by the parent/primary caregiver over the previous month on a 7-point Likert scale (0 = Never, 6 = Always). Items are summed to create total frequency scores for each subscale.
Change in frequency of dysfunctional parenting | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Dysfunctional parenting behavior will be assessed using the Arnold Parenting Overreactivity subscale (PS, 10 items), which examines parent attitudes and beliefs regarding authoritarian discipline. PS responses are based on a 7-point Likert scale in which parents are presented with a situation and then are given two opposing responses at either side of the scale, with the mid-point representing neither one way or the other and the three points on either side of the mid-point representing "sometimes," "generally," and "very often" as one moves further out from the middle. One such item under this subscale is "When my child misbehaves, I raise my voice or yell…I speak to my child calmly." (7 = I raise my voice or yell; 1 = I speak to my child calmly.) Scoring for this subscale is computed by averaging the responses on these items.
Change in frequency of child monitoring and supervision practices | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Parental monitoring and supervision practices will be measured using an adapted version of the Alabama Parenting Questionnaire (APQ) Poor Monitoring/Supervision subscale (11 items). The APQ measures parenting characteristics that have been associated with disruptive behaviour disorders in school-age children, although it has also been used with preschool children. The Poor Monitoring/Supervision subscale will be used to measure the frequency of negative parent monitoring and supervision practices over the past month through a 5-point Likert scale (0 = Never; 5 = Always). Items include "Does (the target child) stay out later than he/she is supposed to?" and "Is (the target child) left at home without adult supervision?" The items in the scale are summed to obtain a total scale score.
Change in frequency of child neglect | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Child neglect will be assessed using an adapted version of the ICAST-T Caregiver tool (mentioned above) Neglect subscale. This subscale has 6 items for assessing medical, physical, and educational neglect, including "In the past month, how often was [Child Nickname] not taken care of when sick or injured, even when you or another caregiver were able to do so and could afford it?" and "In the past month, how often was [Child Nickname] not given a meal that he or she needed, even when you or another caregiver was able to afford it?"
Change in levels of parental depression, anxiety and stress | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Parental depression, anxiety, and stress will be assessed through the Depression, Anxiety, and Stress Scale short form (DASS-21) (21 items) . The DASS-21 will assess parent/primary caregiver depression and anxiety using a 4-point Likert scale [0= Never; 3 = Always] to measure the frequency of symptoms over the previous week. Items include statements such as "I felt that I had nothing to look forward to." Total DASS scores range from 0 to 63, with subscales from 0 to 21. The recommended cut-offs that indicate severity of depression are 5-6 (mild), 7-10 (moderate), 11-13 (severe), and 14 and up (extremely severe), while cut-offs for anxiety are 4-5 (mild), 6-7 (moderate), 8-9 (severe), and 10 and up (extremely severe). Cut-offs for stress are 8-9 (mild), 10-12 (moderate), 13-16 for (severe), and 17 and up (extremely severe).
Change in frequency of child behaviour problems | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  For the purpose of assessing child behaviour problems by parent/primary caregiver self-report, the study will utilize the Eyberg Child Behaviour Inventory (ECBI) Intensity Scale and Problem Scale (36 items). The Intensity Scale measures the frequency of child externalizing behaviours over the past month, using a 7-point Likert-like scale (1 = Never occurs; 7 = Always occurs). Both scales are summed to create a total Intensity Score and Problem Score, with clinical cut-off scores for disruptive behaviour problems suggested as 131 for the Intensity Score and 15 for the Problem Score in the USA. However, no Thai norms are available.
Change in attitudes toward punishment | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Attitudes toward punishment will be assessed using one item from the UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline module. The MICS item asks the parent/primary caregiver: "In order to bring up, raise up, or educate a child properly, the child needs to be physically punished." Parents/primary caregivers will report whether they disagree or agree with the statement based on a 5-point Likert scale of 0 to 4 (0 = Disagree strongly; 4 = Agree strongly).
Change in number of daily child behaviour problems and parenting behaviors | T1: baseline; T2: 1 month; T2: 2 months; T3: 3 months; T4: 6 months
  An adapted version of the Parent Daily Report Checklist (PDR, 44 items) will be used to assess day-to-day occurrences of child behaviour problems and parenting behaviour. In order to assess child behaviour, the PDR asks parents/primary caregivers whether a child externalizing behaviour (e.g. destructiveness, lying, hitting others) occurred within the previous 24 hours (34 items), as well as how much sleep the child had (1 item). To assess parenting behaviour, the PDR asks parents about their own behaviour (6 items, e.g. yelled or shouted at the child, praised child for doing something well) and self-efficacy (3 items, e.g. had a feeling that I could not cope with parenting). Responses to these items are dichotomous (0 = No; 1 = Yes), with items summed for each subscale on parent and child behaviour. The item regarding sleep is a numerical response.
Change in number of positive parent-child interactions | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Parent-child relationships will be measured through a combination of interview and observational items (27 in total), using a combined and adapted version of the Early Childhood and Middle Childhood HOME Inventory record forms, as aforementioned. The HOME Inventory is scored dichotomously. The adapted version contains 16 items on the "responsivity" sub-scale; 6 relevant items on the "encouragement of maturity" sub-scale; 2 items on the "emotional climate" sub-scale; and 2 items on the "modelling" sub-scale.
Change in frequency of Intimate partner violence | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Adult self-report of experiencing intimate partner violence over the past month will be assessed using an adapted version of the Revised Conflict Tactics Scale Short Form (CTS2S, 6 items). This scale includes 2 items on the frequency of negotiation (e.g., "partner suggested a compromise for a disagreement"), 5 items on physical assault (e.g., "partner pushed, shoved, or slapped me"), and 1 item on psychological aggression (e.g., "partner insulted, shouted, yelled, or swore at me"). Answers are coded on a frequency scale of 0 to 3 (0 = never happened; 1 = once or twice; 2 = 3-5 times; 3 = More than 5 times). The CTS2S will determine an overall indication of intimate partner violence on a level of severity (sum of items) and prevalence (dichotomous variable indicating experience of conflict or not), as well as for each subscale.
Change in frequency of attitudes towards corporal punishment | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Adult report of ICAST-T Attitudes subscale (4 items). These items concern a hypothetical scenario of a child with behavioral problems, and parents report whether different disciplinary methods (e.g., "hitting or spanking the child") were effective or ineffective according to a 5-point Likert scale. Items are summed.
Change in frequency of parental sense of inefficacy | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Parent sense of inefficacy will be assessed using an adapted version of the ICAST-Trial Inefficacy Subscale (2 items, e.g., "In the past month, how often did you not know what to do when your child misbehaved?") The items are summed for a total score ranging from 0 to 16 with higher scores indicating a greater sense of inefficacy in managing difficult child behaviour.
Change in frequency of intimate partner coercion | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Adult report of partner coercion based on the WHO questionnaire on women's health and life events (10 items) (Garcia-Moreno, Jansen, Ellsberg, Heise, & Watts, 2005). The WHO assesses experiences of partner coercion (e.g., "partner took your earnings or savings from you against your will"). Responses are scored on a frequency scale of 0-8, with items for each instrument summed to obtain a total score, as well as a score for the negotiation subscale.
Change in frequency of intimate partner negotiation | Differences between groups at T2 (4 months) and T3 (7 months), controlling for T1 (baseline)
  Adult report of Intimate partner violence (IPV) negotiation (2 items; e.g., "partner suggested a compromise for a disagreement"). Items are summed.

OTHER OUTCOMES:
Implementation fidelity | This outcome measure will be assessed once per week over an 8 week period, during parenting programme delivery.
  Fidelity of programme implementation will be measured via self-report checklists by facilitators (Appendix F). The self-report checklist will gauge the level of adherence to the Facilitator Manual, and will include specific activities that the facilitator must deliver for each of the weekly sessions, such as home practice discussions and role-playing exercises.
Implementation quality | The outcome measure will be assessed twice during the 8 week period of parenting programme delivery, during week 6 and week 7.
  Quality of delivery will be assessed by coaches observing the delivery of programme sessions six and seven (two sessions per facilitator) using the Parenting for Lifelong Health Facilitator Assessment Tool (PLH-FAT). The PLH-FAT, similar to the Leader Observation Tool for the Incredible Years parenting programme, is an observational treatment fidelity tool used to assess the process skills necessary for delivery of the programme. It will examine whether and to what extent core intervention components have been delivered, including questions regarding topics touched on per session, such as home practice discussion and role-playing activities. Seven standard behaviour categories are grouped into two scales based on the core activities (23 items) and process skills (28 items) as outlined in the programme manual.
Adherence/exposure (parents/primary caregivers) | This outcome measure will be assessed once per week over an 8 week period, during parenting programme delivery.
  For the purpose of measuring adherence and exposure to the parenting programme, attendance registers will be kept for each weekly session in order to assess the level of exposure of participants to the intervention components.
Engagement in home activities | This outcome measure will be assessed once per week over an 8 week period, during parenting programme delivery.
  Participant engagement in home activities will be measured through weekly participant self-reports of home activity completion, using parent home practice checklists (Appendix H). Participants will complete the forms on a daily basis following the first seven weekly sessions, and these will be collected by facilitators at the beginning of sessions two through eight and maintained in participant case profiles. The forms will indicate to what extent the participants were able to practice the home activities assigned during the previous week's session and in accordance with the intervention manual.
Satisfaction/acceptability/engagement: quantitative data (parents/primary caregivers) | Quantitative data on engagement & acceptability will be assessed once per week over 8 weeks during programme delivery. Quantitative data on satisfaction will be assessed 7 months post-baseline.
  Quantitative data on participant satisfaction will be assessed through a satisfaction questionnaire (45 items) that will be administered to post-intervention, adapted from questionnaires used to evaluate PLH for Young Children programmes during RCTs in South Africa and the Philippines.
  Quantitative data concerning participant engagement and programme acceptability will also be assessed through participant case profiles, which are maintained by facilitators on a weekly basis and will contain notes regarding how individual participants react or engage with the programme material.
Satisfaction/acceptability (facilitators and coaches) | Once per week over 8 weeks during programme delivery, and at T: 7 months
  Qualitative data on facilitator and coach satisfaction/acceptability of the programme will be gathered via a focus group discussion with all facilitators and coaches following programme conclusion.
  Data will also be captured through facilitator session reports and coaching reports. Facilitator session reports will include descriptions of their positive and negative experiences in delivering the programme material. Coaching reports will consist of information from weekly coaching sessions on their coaching experiences, including approaches or issues that worked particularly well or challenging areas that required further attention.
Programme engagement | Baseline
  During the feasibility pilot, obstacles to programme engagement for participants will be assessed using the Obstacles to Engagement Scale (OES) (15 items). The OES measures the influence of personal and intervention-based obstacles to attending the parenting programme sessions. The scales asks parents/primary caregivers to rate each item on a 4-point scale (1=Definitely no; 4 = Definitely yes), with four sub-scales measuring personal or family stressors and obstacles (4 items), relevance of and trust in the intervention (4 items), intervention demands (4 items), and time and scheduling demands (2 items).
Satisfaction/acceptability/engagement: qualitative data (parents/primary caregivers) | Once per week over 8 weeks during programme delivery, and at T: 7 months
  Qualitative data will be gathered through in-depth interviews with 12 parents/primary caregivers, conducted following programme completion. The Interviews will be conducted according to an interview guide, with five broad questions that explore issues of participant satisfaction and perceptions of acceptability according to the themes of: overall programme experience, learning and practicing parenting skills, programme delivery methods, scheduling, and logistics.
  Additional information concerning participant perceptions of engagement and programme acceptability will also be assessed through participant case profiles, which are maintained by facilitators on a weekly basis and will contain notes regarding how individual participants react or engage with the programme material.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Gardner, DPhil, Principal Investigator — University of Oxford; Jamie Lachman, DPhil, Principal Investigator — University of Oxford; Sombat Tapanya, PhD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit; Phaikyeong Cheah, PhD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (4):
- Thailand (4):
  - Ban Tat Health Promotion Hospital, Udon Thani
  - Chiang Pin Health Promotion Hospital, Udon Thani
  - Kling Kam Health Promotion Hospital, Udon Thani
  - Na Phu Health Promotion Hospital, Udon Thani

IPD SHARING:
Plan to Share IPD: Yes
Following the data analyses, all participant data will be de-identified and stored using United Kingdom Data Archive standards (www.data-archive.ac.uk/create-manage/planning-for-sharing). De-identification will include removal of direct identifiers (names, addresses, postcode information, telephone numbers or pictures) as well as indirect identifiers (information on location, occupation or any other information that could be linked to a public source). This will include removing or aggregating variables or reducing the precision or detailed textual meaning of a variable in the dataset. Access to this data will be controlled and require authorisation from the research team for further use.
Supporting Information: Study Protocol
Time Frame: Indefinitely
Access Criteria: Accessibility of the data will require approval from the study team. The study investigators, led by the PI, will jointly make decisions on whether to supply research data to potential new users. Research data will be deposited in and available in the UK Data Archive solely for non-profit use.

REFERENCES:
- [Result] McCoy A, Lachman JM, Ward CL, Tapanya S, Poomchaichote T, Kelly J, Mukaka M, Cheah PY, Gardner F. Feasibility pilot of an adapted parenting program embedded within the Thai public health system. BMC Public Health. 2021 May 29;21(1):1009. doi: 10.1186/s12889-021-11081-4. PMID 34051772
- See also: Parenting for Lifelong Health - Thailand research project page — https://www.spi.ox.ac.uk/parenting-for-lifelong-health-thailand